CLINICAL TRIAL: NCT02740556
Title: Evaluation of HepCure Toolkit to Improve Harvoni Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 15-1273; GS-IN-US-337-3933 (Other Grant/Funding Number: Gilead Sciences)
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Hepatitis C; Medication Adherence
Keywords: Hepatitis C; Adherence; Adheretech; HepCure; Telehealth; Health apps
MeSH Terms: conditions — Hepatitis C; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AdhereTech Passive Monitoring (Placebo Comparator): Patients not using the HepCure patient app while AdhereTech passively monitors adherence (no chimes or reminders).
  Interventions: Other: AdhereTech Passive Monitoring
- HepCure Toolkit (Experimental): Patients using the HepCure patient app linked to a provider using the HepCure Provider Dashboard with AdhereTech passively monitoring adherence (no chimes or reminders).
  Interventions: Other: HepCure ToolKit; Other: AdhereTech Passive Monitoring
- HepCure Toolkit and AdhereTech Active Features (Experimental): Patients using the HepCure patient app linked to a provider using the HepCure Provider Dashboard and with AdhereTech actively monitoring adherence (chimes and reminders enabled).
  Interventions: Other: HepCure ToolKit; Device: AdhereTech Active Features

INTERVENTIONS:
Other: HepCure ToolKit — HepCure is a web-based tool kit in the form of a dashboard for providers and an application (or "app") for patients. The app allows patients to become active participants in their treatment by enabling them to enter prescribed treatment, add medications to "Pill Box," log doses, visualize adherence, and includes several additional resources.
  Arms: HepCure Toolkit; HepCure Toolkit and AdhereTech Active Features
Device: AdhereTech Active Features — AdhereTech, a wireless pill monitoring device that measures the dosage and time a medication was taken. It is a HIPAA-compliant, FDA-registered Class I medical device. Using cellular technology, AdhereTech can be used passively to collect data on when a medication is taken, when a refill is needed, and how often the bottle is opened. AdhereTech also can be used actively to monitor adherence and provide feedback to subjects using the device. When actively monitoring, AdhereTech can be set up to provide live feedback to a subject by lighting up, sounding chimes, and sending phone/text/email alerts to remind patients to take their medication.
  Arms: HepCure Toolkit and AdhereTech Active Features
Other: AdhereTech Passive Monitoring — AdhereTech passively monitors adherence (no chimes or reminders)
  Arms: AdhereTech Passive Monitoring; HepCure Toolkit

SUMMARY:
There is limited data outside of clinical trials on adherence to once daily ledipasvir/sofosbuvir regimens. Many patients present with known barriers to medication adherence including untreated psychiatric illness and substance use disorders, cognitive impairment, and low health literacy. The goal of this study is to evaluate the baseline level of adherence to ledipasvir/sofosbuvir in a real-world clinic population and compare this to the level of adherence in patients provided with additional adherence support. Medication adherence in this study will be evaluated using AdhereTech, a wireless pill monitoring device that measures the dosage and time a medication was taken. Using cellular technology, AdhereTech can be used passively to collect data on when a medication is taken, when a refill is needed, and how often the bottle is opened. AdhereTech also can be used actively to monitor adherence and provide feedback to subjects using the device. When actively monitoring, AdhereTech can be set up to provide live feedback to a subject by lighting up, sounding chimes, and sending phone/text/email alerts to remind patients to take their medication (see attached PowerPoint presentation). HepCure is a web-based tool kit in the form of a dashboard for medical providers (MDs and NPs) and an application (or "app") for patients. The app allows patients to become active participants in their treatment by enabling them to set medication reminders, record doses taken, and communicate their adherence to their medical provider using the provider dashboard.

DETAILED DESCRIPTION:
Primary Objectives:

The study will be conducted in two phases with the following aims: (1) To passively assess the adherence to hepatitis C virus (HCV) treatment with ledipasvir/sofosbuvir using a wireless pill monitoring device in 33 patients (Phase 1, months 1-3). (2) To test the impact on adherence of using the active wireless pill monitoring device in conjunction with the HepCure web-based tool kit in 66 patients (Phase 2, months 4-9). Participants in phase 2 will be randomized 1:1 to one of two conditions: (a) Patients using the HepCure patient app linked to a provider using the HepCure Provider Dashboard; AdhereTech passively monitoring adherence. (b) Patients using the HepCure patient app linked to a provider using the HepCure Provider Dashboard; AdhereTech actively monitoring adherence (chimes and reminders enabled).

Secondary Objectives:

The study design allows us to compare the additive effect on adherence of the HepCure provider toolkit and the HepCure provider toolkit + active AdhereTech reminder system.

Primary Endpoints:

The primary study endpoints are taking and timing adherence as assessed by electronic monitoring. There are numerous methods of assessing adherence to medication. They each have their strengths and weaknesses, and some are only feasible in the research but not clinical setting. The most commonly used methods of assessing adherence are (1) provider assessment, (2) structured self-report (3) pharmacy refill data (4) electronic monitoring (5) pill counts and (6) directly observed therapy. Electronic monitoring technology has been widely used in research studies of HIV medication adherence and is regarded by many as the most accurate method of assessing medication adherence (Weiss et al. 2009). In this method, the medication bottle cap has a microchip which records all openings and closings of the bottle. This microchip provides the researcher with a precise record of the date and time of each bottle opening. This method has been shown to be closely associated with random home pill count (Bangsberg et al., 2001a), viral suppression (Bangsberg et al., 2000; Paterson et al., 2000; Arnsten et al., 2001; Walsh et al., 2002b; Moss et al., 2004), and drug resistance (Walsh et al., 2002b). Studies have consistently found that provider assessment of adherence is poor (Bangsberg et al., 2001b; Gross et al., 2002; and Miller et al., 2002). Self-reported adherence tends to provide an over-estimate of actual adherence (Weiss et al. 2009). Pharmacy refill data is best employed when patients use one pharmacy for all prescriptions, pharmacy data are easily accessible to the clinician by computer, and prescriptions are not automatically delivered without the patient needing to request them or pick them up. Patients in clinical research studies are often asked to bring their medication to study visits so that the change in the number of pills (accounting for refills) since the last visit can be used to assess adherence. Potential problems associated with these announced pill counts are that patients may forget to bring their medication to study visits, and nonadherent patients may throw out pills prior to the visit ("pill dumps") to avoid being labeled nonadherent. While directly observed therapy (DOT) provides a highly accurate assessment of adherence, the cost and intrusiveness of observing all doses of medication ingestion make it an impractical method of ARV adherence assessment, except in very specific settings (e.g., prisons or nursing homes).

ELIGIBILITY:
No one will be excluded based on gender, age, race, or ethnic group.

Inclusion criteria Phase 1 and 2:

* Age18 years and older
* Being prescribed Harvoni for treatment of HCV and not yet started treatment
* Speak and read English

Inclusion criteria Phase 2 Only:

* Possessing a smartphone device
* Ability to use a smartphone device
* Registered with a physician currently using the HepCure Provider Dashboard.
* Speak and read English

Exclusion criteria:

* Individuals with diminished mental capacity who are unable to give informed consent
* Prisoners
* Participants who do not speak or write in English as a primary language
* Participants who are unable to speak and read English
* Participants who are expected to have difficult with regular access to smart phone device.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-02; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | up to 9 months
  AdhereTech bottles use sensors to provide a timestamp of when the bottle cap was open and closed.

SECONDARY OUTCOMES:
HCV RNA | up to 9 months
  The Sustained Viral Response (SVR) outcome will be monitored until the patient attains sustained virologic response post-treatment measured by HCV RNA from medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Weiss, PhD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnsten JH, Demas PA, Farzadegan H, Grant RW, Gourevitch MN, Chang CJ, Buono D, Eckholdt H, Howard AA, Schoenbaum EE. Antiretroviral therapy adherence and viral suppression in HIV-infected drug users: comparison of self-report and electronic monitoring. Clin Infect Dis. 2001 Oct 15;33(8):1417-23. doi: 10.1086/323201. Epub 2001 Sep 5. PMID 11550118
- [Background] Bangsberg DR, Hecht FM, Charlebois ED, Zolopa AR, Holodniy M, Sheiner L, Bamberger JD, Chesney MA, Moss A. Adherence to protease inhibitors, HIV-1 viral load, and development of drug resistance in an indigent population. AIDS. 2000 Mar 10;14(4):357-66. doi: 10.1097/00002030-200003100-00008. PMID 10770537
- [Background] Bangsberg DR, Hecht FM, Charlebois E, Chesney M, and Moss AR (2001a). Comparing objective methods of adherence assessment: electronic medication monitoring and unannounced pill count. AIDS Behav 5:275-281.
- [Background] Bangsberg DR, Perry S, Charlebois ED, Clark RA, Roberston M, Zolopa AR, Moss A. Non-adherence to highly active antiretroviral therapy predicts progression to AIDS. AIDS. 2001 Jun 15;15(9):1181-3. doi: 10.1097/00002030-200106150-00015. No abstract available. PMID 11416722
- [Background] Fennie KP, Bova CA, Williams AB. Adjusting and censoring electronic monitoring device data. Implications for study outcomes. J Acquir Immune Defic Syndr. 2006 Dec 1;43 Suppl 1:S88-95. doi: 10.1097/01.qai.0000248336.97814.2f. PMID 17133208
- [Background] Gross R, Bilker WB, Friedman HM, Coyne JC, Strom BL. Provider inaccuracy in assessing adherence and outcomes with newly initiated antiretroviral therapy. AIDS. 2002 Sep 6;16(13):1835-7. doi: 10.1097/00002030-200209060-00021. PMID 12218400
- [Background] Miller LG, Liu H, Hays RD, Golin CE, Beck CK, Asch SM, Ma Y, Kaplan AH, Wenger NS. How well do clinicians estimate patients' adherence to combination antiretroviral therapy? J Gen Intern Med. 2002 Jan;17(1):1-11. doi: 10.1046/j.1525-1497.2002.09004.x. PMID 11903770
- [Background] Moss AR, Hahn JA, Perry S, Charlebois ED, Guzman D, Clark RA, Bangsberg DR. Adherence to highly active antiretroviral therapy in the homeless population in San Francisco: a prospective study. Clin Infect Dis. 2004 Oct 15;39(8):1190-8. doi: 10.1086/424008. Epub 2004 Sep 27. PMID 15486844
- [Background] Paterson DL, Swindells S, Mohr J, Brester M, Vergis EN, Squier C, Wagener MM, Singh N. Adherence to protease inhibitor therapy and outcomes in patients with HIV infection. Ann Intern Med. 2000 Jul 4;133(1):21-30. doi: 10.7326/0003-4819-133-1-200007040-00004. PMID 10877736
- [Background] Walsh JC, Pozniak AL, Nelson MR, Mandalia S, Gazzard BG. Virologic rebound on HAART in the context of low treatment adherence is associated with a low prevalence of antiretroviral drug resistance. J Acquir Immune Defic Syndr. 2002 Jul 1;30(3):278-87. doi: 10.1097/00126334-200207010-00003. PMID 12131564
- [Background] Weiss JJ, Brau N, Stivala A, Swan T, Fishbein D. Review article: adherence to medication for chronic hepatitis C - building on the model of human immunodeficiency virus antiretroviral adherence research. Aliment Pharmacol Ther. 2009 Jul;30(1):14-27. doi: 10.1111/j.1365-2036.2009.04004.x. Epub 2009 Mar 26. PMID 19416131